CLINICAL TRIAL: NCT00230295
Title: Indirect Magnetic Resonance Lymphangiography of the Head and Neck Region Using Conventional Gadolinium-based Contrast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Quynh-Thu Le, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENT0010; ENT0010; NCT00230295
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Head and Neck Cancer; Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms

INTERVENTIONS:
Procedure: IMR LAG

SUMMARY:
To determine the ability of magnetic resonance lymphangiography using conventional gadolinium injected directly into the tumor site and PET scan in detecting microscopic nodal metastasis in patients with newly diagnosed H&N cancers

ELIGIBILITY:
Inclusion Criteria:Patients with newly diagnosed squamous cell carcinomas of the H&N with primary tumor sites that are accessible to direct contrast injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determined the ability of magnetic resonance lymphangiography using conventional gadolinium injected directly into the tumor site and PET scan in detecting microscopic nodal metastasis in patients with newly diagnosed H&N cancers

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States